CLINICAL TRIAL: NCT04128501
Title: A Phase II Study of Venetoclax in Combination With Azacitidine in the Post-Transplant Setting for AML, T Cell Leukemia, and Mixed Phenotype Acute Leukemia
Brief Title: Venetoclax and Azacitidine for the Treatment of Acute Myeloid Leukemia in the Post-Transplant Setting
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0353; NCI-2019-06674 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0353 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Acute Bilineal Leukemia; Acute Biphenotypic Leukemia; Acute Myeloid Leukemia; Mixed Phenotype Acute Leukemia; T Acute Lymphoblastic Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, venetoclax) (Experimental): Patients receiving venetoclax and azacitidine for maintenance after allogeneic stem cell transplantation, receive azacitidine SC on days 1-5 and venetoclax PO QD on days 1-7. Patients receiving venetoclax and azacitidine for minimal residual disease after allogeneic stem cell transplant, receive azacitidine SC on days 1-5 and venetoclax PO QD on days 1-14. Treatment repeats every 4-8 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well venetoclax and azacitidine work for the treatment of acute myeloid leukemia after stem cell transplantation. Venetoclax may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax and azacitidine after a stem cell transplant may help control high risk leukemia and prevent it from coming back after the transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. To determine relapse-free survival after the use of venetoclax in combination with azacitidine given as maintenance therapy or for eradication of minimal residual disease in patients with high risk acute myeloid leukemia (AML) after hematopoietic stem cell transplantation (HSCT).

SECONDARY OBJECTIVES:

1. To determine the safety and toxicity of venetoclax in combination with azacitidine (type, frequency, severity of adverse events [AEs] and relationship of AEs to venetoclax)
2. To determine response duration, overall survival.
3. To determine Incidence of acute and chronic graft versus host disease (GVHD)
4. To perform matched pairs analysis to obtain bias corrected treatment comparisons of Venetoclax + Vidaza (V+V) to standard therapy in AML patients with no evidence of disease (AML D-) subgroup.

EXPLORATORY OBJECTIVE:

1. To investigate possible relationships between baseline protein and gene expression signatures/mutation profile and BH3 profiling in predicting relapse-free survival time to the combination. This exploratory analysis will be done for the data from the entire study, accounting for the noted biological variables covariates, as well as disease status and whether or not the patient had AML, by fitting a Bayesian time-to-event regression model with RFS the outcome variable.

OUTLINE:

Patients receiving venetoclax and azacitidine for maintenance after allogeneic stem cell transplantation, receive azacitidine subcutaneously (SC) on days 1-5 and venetoclax orally (PO) once daily (QD) on days 1-7. Patients receiving venetoclax and azacitidine for minimal residual disease after allogeneic stem cell transplant, receive azacitidine SC on days 1-7 and venetoclax PO QD on days 1-14. Treatment repeats every 4-8 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 18 to 75 years of age.
2. English and non-English speaking patients are eligible.
3. Disease diagnosis with one of the hematological malignancies listed below and who are in morphological remission after allogeneic stem cell transplantation with PBSCs or bone marrow.

   1. AML if they had at least one of the following disease characteristics:

      * Therapy related AML.
      * Cytogenetics and molecular features consistent with adverse risk group by European LeukemiaNet classification for AML (see Appendix A.).
      * Primary induction failure defined as absence of complete remission after two different lines of anti-leukemia therapy following diagnosis.
      * Presence of minimal residual disease by multi-color flow cytometry or cytogenetics or molecular studies at the time of HSCT.
      * Presence of active disease defined as bone marrow blast count >5% at the time of HSCT.
      * Participants transplanted beyond first remission. OR
   2. Biphenotypic or bilineage leukemia (including a myeloid component) OR mixed phenotype acute leukemia (MPAL) OR
   3. Participants with acute lymphoblastic leukemia; B cell or T cell in original.
4. Participants in morphological remission with no detectable minimal residual disase (MRD) after transplant
5. Participants who are in remission with no detectable minimal residual disease (MRD) after allogeneic stem cell transplant should have:

   1. Adequate engraftment within 14 days prior to starting study drug:
   2. Absolute neutrophil count (ANC) >/= 1.0 x 109/L without daily use of myeloid growth factor (G-CSF) for at least 7 days; and,
   3. Platelet >/= 30 x 109/L without platelet transfusion within 1 week
   4. Be able to start the drug therapy between 42 to 100 days following HSCT.
6. Use of one of the conditioning regimens as part of allogeneic stem cell transplant listed below:

   1. Reduced intensity regimen with fludarabine/melphalan (100-140 mg/m2) with or without TBI with post-transplant Cytoxan OR
   2. Myeloablative regimens including:

      * Busulfan (AUC at or greater than 4000)/fludarabine with post-transplant Cytoxan or total body irradiation (TBI)/etoposide with any graft versus host disease (GVHD) regimen OR
      * Total body irradiation (TBI)/etoposide with any graft versus host disease (GVHD) regimen.
7. Participants on clinical trials investigating different conditioning regimens (with the above described backbone) with investigational agents will be allowed to enroll.
8. ECOG performance status of 0, 1, or 2.
9. Serum creatinine </=1.5 mg/dL or creatinine clearance greater or equal than 40 cc/min as defined by the Cockcroft-Gault Equation*
10. Serum bilirubin </= 1.5 x upper limit of normal (ULN).
11. Aspartate transaminase (AST) or alanine transaminase (ALT) </= 2.5 x ULN.
12. Alkaline phosphatase </= 2.5 x UL.
13. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
14. Negative serum or urine pregnancy test for women with reproductive potential. The only subjects who will be exempt from this criterion are postmenopausal women (defined as women who have been amenorrheic for > 12 months) or subjects who have been surgically sterilized or otherwise proven sterile. 3.1.2. For cohort #3 and cohort #4 patients (MRD positive cohort):

<!-- -->

1. Participants 18 to 75 years of age.
2. English and non-English speaking patients are eligible.
3. Disease diagnosis with one of the hematological malignancies listed below and who are in morphological remission after allogeneic stem cell transplantation with PBSCs or bone marrow. a. AML OR b. Biphenotypic or bilineage leukemia (including a myeloid component) or mixed phenotype acute leukemia (MPAL) OR c. Participants with acute lymphoblastic leukemia; B cell or T cell in original.
4. Persistence or reappearance of MRD by flow cytometry or cytogenetic or molecular testing while being in morphological remission after allogeneic stem cell transplantation.

   1. When MRD is detected by flow cytometry, disease level at or above the sensitivity level of the test will be required. • MRD level at or above 0.01% for B cell ALL and T cell ALL.

      • MRD level at or above 0.1% for AML and mixed phenotype acute leukemia.
   2. When MRD is detected by cytogenetics, disease level at or above the sensitivity level of the test will be required.

      • The limited of detection is about 0.25% for males and 0.44% for females.
   3. When MRD is detected by molecular testing, disease level at or above the sensitivity level of the test will be required. • The limited of detection is 0.01%
5. Use of one of the conditioning regimens as part of allogeneic stem cell transplant listed below:

   a. Reduced intensity regimen with fludarabine/melphalan (100-140 mg/m2) with or without TBI with post-transplant Cytoxan OR b. Myeloablative regimens including:

   • Busulfan (AUC at or greater than 4000)/fludarabine with post-transplant Cytoxan or total body irradiation (TBI)/etoposide with any graft versus host disease (GVHD) regimen OR
   * Total body irradiation (TBI)/etoposide with any graft versus host disease (GVHD) regimen.
6. Participants on clinical trials investigating different conditioning regimens (with the above described backbone) with investigational agents will be allowed to enroll.
7. ECOG performance status of 0, 1, or 2.
8. Serum creatinine </=1.5 mg/dL or creatinine clearance greater or equal than 40 cc/min as defined by the Cockcroft-Gault Equation*
9. Serum bilirubin </= 1.5 x upper limit of normal (ULN).
10. Aspartate transaminase (AST) or alanine transaminase (ALT) </= 2.5 x ULN.
11. Alkaline phosphatase </= 2.5 x UL.
12. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
13. Negative serum or urine pregnancy test for women with reproductive potential. The only participants who will be exempt from this criterion are postmenopausal women (defined as women who have been amenorrheic for > 12 months) or subjects who have been surgically sterilized or otherwise proven sterile.

Exclusion Criteria:

1. Active acute GVHD grade II or higher.
2. Active chronic GVHD that is extensive (see Appendix C.).
3. Uncontrolled GVHD (see Appendix C.).
4. Concurrent use of systemic immune suppressive other than calcineurin inhibitors, sirolimus and steroids
5. Active uncontrolled systemic fungal, bacterial or viral infection.
6. Active bleeding.
7. Symptomatic or uncontrolled arrhythmias.
8. Significant active cardiac disease within the previous 6 months, including:

   1. New York Heart Association (NYHA) class III or IV congestive heart failure see Appendix C.).

   Unstable angina or angina requiring surgical or medical intervention, and/or b. Myocardial infarction.
9. Known active viral infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV).
10. Prior history of malignancies, other than leukemia, unless the subject has been free of the disease for >/= 1 year. However, participants with the following history/concurrent conditions are allowed:

    1. Basal or squamous cell carcinoma of the skin;
    2. Carcinoma in situ of the cervix;
    3. Carcinoma in situ of the breast;
    4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis [TNM] clinical staging system).
11. Participants with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) time | From the date of first administration of venetoclax + azacitidine (vidaza) (V+V), assessed up to 60 days after last V+V dose
  Summary statistics for RFS time will be computed for all patients and within each (disease status, disease type) subgroup. RFS time distributions will be estimated within each subgroup using the method of Kaplan and Meier.

SECONDARY OUTCOMES:
Overall survival (OS) time | Up to 60 days after last V+V dose
  Summary statistics for OS time will be computed for all patients and within each (disease status, disease type) subgroup. OS time distributions will be estimated within each subgroup using the method of Kaplan and Meier.
Incidence of severe (grade 3 or 4) infection | Up to 60 days after last V+V dose
  Will be summarized, and relevant parameters will be estimated under appropriate Bayesian models.
Graft-versus-host disease | Up to 60 days after last V+V dose
  Will be summarized, and relevant parameters will be estimated under appropriate Bayesian models.
Incidence of other inter-current adverse events during follow up | Up to 60 days after last V+V dose
  Will be summarized, and relevant parameters will be estimated under appropriate Bayesian models.
Non-relapse mortality | Within 90 days from the start of V+V treatment
  Defined as death from any cause, within 90 days from the start of V+V treatment that is not preceded by disease recurrence. Will be summarized, and relevant parameters will be estimated under appropriate Bayesian models.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Oran, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org